CLINICAL TRIAL: NCT00214838
Title: An Open-Label Study of the Safety and Efficacy of Atiprimod Treatment for Patients With Advanced Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Callisto Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-102
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2006-12-05 (Estimated); Status verified 2006-12

CONDITIONS: Advanced Cancer
Keywords: cancer, atiprimod
MeSH Terms: conditions — Neoplasms | interventions — azaspirane

INTERVENTIONS:
Drug: Atiprimod

SUMMARY:
The primary objectives of this study are to identify the maximum tolerated dose and to evaluate safety of atiprimod in patients with advanced cancer.

DETAILED DESCRIPTION:
The primary objectives of this study are to identify the maximum tolerated dose(MTD) and to evaluate safety of atiprimod in patients with advanced cancer.

The secondary objectives of this study are 1) to measure the pharmacokinetics of atiprimod and 2) to evaluate the efficacy of atiprimod treatment in patients with advanced cancers and 3) to compare the pharmacokinetics of atiprimod tablets and capsules at the starting dose, with the intent of switching to capsules for the dose escalation if the capsules pose no safety issues.

ELIGIBILITY:
Inclusion Criteria:

* histological proof of advanced cancer and must have failed or relapsed following standard therapy or have no standard therapy available.
* estimated life expectancy of at least 12 weeks.
* must have evaluable disease.
* ECOG(Zubrod) PS of 0 to 2
* sign informed consent.
* age 13 years or more at time of signing informed consent.

Exclusion Criteria:

* renal insufficiency
* concomitant radiotherapy, chemotherapy or other investigational therapies.
* peripheral neuropathy grade 3 or greater (NCI CTC version 3 grading)
* evidence of clinically significant mucosal or internal bleeding
* any condition that in the opinion of the investigator, places the patient at unacceptable risk if he/she were to participate in the study.
* clinically relevant active infection or serious co-morbid medical conditions.
* as atiprimod is a potent inhibitor of CYP2D6, patients taking drugs that are substrates of CYP2D6(e.g. beta blockers, antidepressants and antipsychotics will be excluded.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61
Dates: Start 2005-03; Study Completion 2007-03

PRIMARY OUTCOMES:
The primary objectives of this study are to identify the maximum tolerated dose
MTD) and to evaluate the safety of atiprimod when given in doses starting at
60 mg/day and ranging to 360 mg/day, or the MTD, whichever is lower, in
patients with advanced cancer.

SECONDARY OUTCOMES:
The secondary objectives of this study are to measure the pharmacokinetics of
atiprimod, to evaluate the efficacy of atiprimod treatment in patients with
advanced cancer, and to compare the pharmacokinetics of atiprimod tablets and
capsules at the starting dose, with the intent of switching to capsules for
the dose escalation if the capsules pose no safety issues.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Picker, PhD, Study Director — Callisto Pharmaceuticals Inc
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States